CLINICAL TRIAL: NCT02731014
Title: Dry Needling for Patients With Neck Pain: A Randomized Clinical Trial
Brief Title: Dry Needling for Patients With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franklin Pierce University (Other)
Collaborators: Newcastle University (Other); Concord Hospital (Other)
Responsible Party: Principal Investigator, Joshua Cleland, DPT, OCS, Professor of Physical Therapy, Franklin Pierce University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIC 15-6
Record Dates: First submitted 2016-03-23; First posted 2016-04-07 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Neck Pain
Keywords: Dry Needling
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Dry Needling Group (Experimental): Dry Needling, Manual Therapy, and Exercise.
  Interventions: Other: Dry Needling; Other: Manual Therapy; Other: Exercise
- Sham Dry Needling Group (Sham Comparator): Sham Dry Needling, Manual Therapy, and Exercise.
  Interventions: Other: Sham Dry Needling; Other: Manual Therapy; Other: Exercise

INTERVENTIONS:
Other: Dry Needling — Dry Needling targeting the posterior musculature of the cervical and thoracic spine.
  Arms: Dry Needling Group
Other: Sham Dry Needling — Sham Dry Needling performed with Park sham acupuncture needles (Acuprime, UK) will be used to perform sham dry-needling. The device consists of 2 plastic tubes that slide into one another and cause a pricking sensation when pushed against the skin.
  Arms: Sham Dry Needling Group
Other: Manual Therapy — Manual Therapy(mobilization/ manipulation) to address joint mobility of the cervical and thoracic spine.
Other: Exercise — Exercise designed to improve performance of both the deep neck flexor musculature as well as the scapular musculature. The exercise portion will also include a stretching program targeting the cervicothoracic muscles which have been placed in a shortened position as a result of poor postures.

SUMMARY:
The aim of this trial will be to examine the short and long term effectiveness of dry needling on pain, disability, and patient perceived improvements in patients with neck pain attending physical therapy. The investigators hypothesize that patients who receive dry needling, manual therapy, and exercise will achieve greater reductions in pain and disability in the short (4 weeks) and long term (6 and 12 months) compared to those who receive sham dry needling, manual therapy, and exercise.

DETAILED DESCRIPTION:
Background: Neck pain is a costly and common problem. Current treatments are not adequately effective for a large proportion of patients who continue to experience recurrent pain. Therefore, new treatment strategies should be investigated in an attempt to reduce the disability and high costs associated with neck pain.

Dry needling is a technique in which a fine needle is used to penetrate the skin, subcutaneous tissues, and muscle with the intent to mechanically disrupt tissue without the use of an anesthetic. Dry needling is emerging as a treatment modality that is widely used clinically to address a variety of musculoskeletal conditions. Recent studies of dry needling in mechanical neck pain have shown decreased pain, increased pain pressure threshold, improved range of motion, and decreased disability in the short term. The majority of these studies examined dry needling using methods atypical to clinical practice (dry needling as a sole treatment, or fewer visits than is common practice). None included long-term follow up. A clinical trial with realistic treatment time frames and methods consistent with clinical practice is needed to examine the effectiveness of dry needling on reducing pain and enhancing function in patients presenting with mechanical neck pain.

Purpose: The aim of this trial will be to examine the short and long term effectiveness of dry needling on pain, disability, and patient perceived improvements in patients with neck pain.

Design: The investigators will conduct a randomized single blind placebo controlled trial in accordance with the CONSORT guidelines. All patients with mechanical neck pain referred to physical therapy will be screened for eligibility criteria. Participants will be randomized to receive 1) dry needling, manual therapy, and exercise or 2) sham dry needling, manual therapy and exercise. Participants will receive 7 treatments over a maximum of 4 weeks.

Methods: The primary outcome will be disability as measured by the Neck Disability Index. Pain and patient perceived improvement will also be recorded. Outcome measures will be assessed at 4 weeks, 6 months, and 12-months by an assessor who is blind to the group allocation of the participants to determine the short and long-term treatment effects.

Data Analysis: The investigators will examine the primary aim with a 2-way repeated-measures analysis of variance (ANOVA) with treatment group as the between subject variable and time as the within-subjects variable. The hypothesis of interest will be the 2-way group by time interaction.

Significance: The successful completion of this trial will provide evidence to demonstrate whether dry needling is effective for the management of mechanical neck pain when used in a combined treatment approach as is commonly practiced clinically.

ELIGIBILITY:
Inclusion Criteria:

1. Age between >18 years old
2. Primary complaint of neck pain
3. Neck Disability Index > 10 points=20%

Exclusion Criteria:

1. Red flags noted in the patient's Neck Medical Screening Questionnaire (i.e. tumor, fracture, metabolic diseases, Rheumatoid Arthritis, osteoporosis, prolonged history of steroid use, symptoms of vertebrobasilar insufficiency, pregnancy, cervical spinal stenosis, bilateral upper extremity symptoms etc.
2. Use of blood thinners
3. History of whiplash injury within the past six weeks
4. Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes), etc.
5. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

   * Muscle weakness involving a major muscle group of the upper extremity
   * Diminished upper extremity muscle stretch reflex (biceps brachii, brachioradialis, or triceps)
   * Diminished or absent sensation to pinprick in any upper extremity dermatome
6. Prior surgery to the neck or thoracic spine
7. Chiropractic, Physical Therapy, or Acupuncture treatment for their neck pain in the last 12-months
8. Workers compensation or pending legal action regarding their neck pain
9. Insufficient English language skills to complete all questionnaires
10. Inability to comply with treatment and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Neck Disability Index (NDI) | 4 weeks, 6 months, 12 months
  The Neck Disability Index (NDI) was created to measure pain related disability associated with activities of daily living in people with neck pain. The NDI contains ten focused sections. The NDI is easy to complete and score. Each item is scored on a 6 point scale and can reach a maximum score of 5; therefore, the maximum score is 50. This score will calculated as a percentage, with higher scores indicating higher levels of disability.

SECONDARY OUTCOMES:
Change from baseline on The Global Rating Of Change Scale (GROC) | 4 weeks, 6 months, 12 months
  The GROC is a 15-point scale used to quantify a patient's improvement with treatment or to record the clinical course of a condition over time. Patients are asked to describe their overall condition since the start of treatment until the present time with options ranging from -7 ("a very great deal worse") to +7 ("a very great deal better") and 0 being described as "about the same."
Questionnaire used to assess blinding of patients to which needling intervention they received | 4 weeks
  Used to assess blinding of patients as to which dry needling intervention the received (real or sham).
Change from baseline on the Visual Analog Scale (VAS) Pain | 4 weeks, 6 months, 12 months
  The VAS is a single item measure of pain using a 100 mm horizontal line anchored on the left side of which represents "no pain" and the right side represents "the worst pain imaginable". The VAS will be used to calculate change in pain score from baseline to 4 weeks, 6 months, and 12 months.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Franciscan, ST.Francis Health, Indianapolis, Indiana
  - Concord Hospital Rehabilitation Services, Concord, New Hampshire

REFERENCES:
- [Derived] Gattie ER, Cleland JA, Snodgrass SJ. Dry Needling for Patients With Neck Pain: Protocol of a Randomized Clinical Trial. JMIR Res Protoc. 2017 Nov 22;6(11):e227. doi: 10.2196/resprot.7980. PMID 29167092